## Randomized Trial to Improve Safe Firearm Storage

NCT05568901

June 1, 2021

Study Name: Firearm Access Reduction Through ER Intervention (FARTHER)

Study Principal Investigator: Mike Gittelman MD

Co-Investigator: Bijan Ketabchi MD, Wendy Pomerantz MD

**Purpose:** Suicide is the #2 cause of death among children. Children with depression, anxiety or other behavioral issues are impulsive and at highest risk for suicide. In this age group, medications are the most common means of attempted suicide, while firearms are the most lethal means of attempted suicide. The purpose of this research study is to identify which methods of counseling and resources are most useful in helping families safely store medications and firearms in order to prevent suicide and unintentional injury among families presenting to the Emergency Room for psychiatric evaluation.

**Procedures:** If you agree to participate, you will be randomized (or assigned) to receive either 1) an information sheet or 2) an information sheet with 2 cable-style firearm locks. You cannot pick which group you are randomized into. Both items are to help you store dangerous items more safely in your own home. Approximately 4 weeks after the visit we will send you a survey link via text that will ask you how you store dangerous items in your home and what your opinion was of the counseling/resources provided to you at this visit.

**Payment:** You will be provided with a \$10 gift card to Target if you agree to participate at this time. You will be sent an additional \$10 Gift Card (either physical card or electronic gift card) after you complete the follow-up survey in 4 weeks. There is no cost to participate in this study.

**Risks:** There are no major risks in participating. There is small risk of loss of confidentiality however, all electronic files will be password protected and only available to research staff for this study.

**Benefits:** The direct benefits to you and your child include resources to help you store dangerous items more safely in order to prevent suicide or accidental injury. With your participation, we hope to identify the optimal information and resources to help our families keep their children safe.

**Your participation is voluntary.** If you choose not to participate, it will not affect your child's care in any way. Answering the survey questions indicates that you agree to participate. If you decide to participate, you can withdraw from the study at any time. Withdrawing from the study also will not affect your child's care in any way.

For questions and concerns regarding this research study you can contact Bijan Ketabchi at (513) 659-6701 or Mike Gittelman at (513) 636-2274. If you have questions regarding your rights as a research participant, then you may contact the Cincinnati Children's Hospital Medical Center Institutional Review Board at (513) 636-8039. Researchers at other sites participating in this study, individuals from the Institutional Review Board (IRB), the Human Subjects Protection Program Office (HSPPO), and other regulatory agencies may inspect these records. In all other respects, however, the data will be held in confidence to the extent permitted by law. Other institutions participating in this research study will not have access to your private health information. Should the data be published, your identity will not be disclosed.